CLINICAL TRIAL: NCT01330134
Title: Comparison of Two Lidocaine Administration Techniques
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10-621A
Record Dates: First submitted 2011-04-04; First posted 2011-04-06 (Estimated); Results first posted 2018-06-28 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-06

CONDITIONS: Pain
Keywords: procedural
MeSH Terms: conditions — Pain | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- lidocaine onto skin prior to lidocaine subcutaneous injection (Experimental): 1-2ml of 1% lidocaine dripped onto the surface of the skin immediately prior to subcutaneous injection of 1% lidocaine.
  Interventions: Drug: lidocaine
- lidocaine subcutaneous injection alone (Active Comparator): 1% lidocaine subcutaneous injection alone by standard approach
  Interventions: Drug: lidocaine

INTERVENTIONS:
Drug: lidocaine — 2ml 1% lidocaine placed onto surface of the skin immediately prior to 1% lidocaine subcutaneous injection
  Arms: lidocaine onto skin prior to lidocaine subcutaneous injection
Drug: lidocaine — 1% lidocaine subcutaneous injection alone
  Arms: lidocaine subcutaneous injection alone

SUMMARY:
The objective of our study is to determine if technique of lidocaine administration can decrease pain perception.

Hypothesis: There will be a significant difference in pain perception between patients who are given lidocaine on the skin surface prior to subcutaneous injection and patients who are given only subcutaneous injection by standard approach.

DETAILED DESCRIPTION:
This is a single center prospective, randomized, blinded study assessing pain perception following 2 different lidocaine administration techniques in subjects who have planned medical procedures requiring local injection of lidocaine. Subjects will be approached and consented to participate in the study. They will be interviewed after the scheduled medical procedure to assess their pain using validated pain scores. An investigator who is not present for the procedure and blinded to the randomization will gather data regarding perceptions of pain from the entire procedure.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients refered to the University of Chicago Medical Centers Procedure Service for a planned medical procedure requiring local injection of lidocaine.

Exclusion Criteria:

* Patient who lack decisional capacity to consent
* Patients who lack the ability to answer questions in english using pain scales

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 481 (Actual)
Dates: Start 2011-02; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John P Kress, MD., Principal Investigator — Univeristy of Chicago
Locations (1):
- The University of Chicago Medical Center, Chicago, Illinois, United States

REFERENCES:
- [Derived] Patel BK, Wendlandt BN, Wolfe KS, Patel SB, Doman ER, Pohlman AS, Hall JB, Kress JP. Comparison of Two Lidocaine Administration Techniques on Perceived Pain From Bedside Procedures: A Randomized Clinical Trial. Chest. 2018 Oct;154(4):773-780. doi: 10.1016/j.chest.2018.04.018. Epub 2018 Apr 24. PMID 29698720

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lidocaine Onto Skin Prior to Lidocaine Subcutaneous Injection | Lidocaine Subcutaneous Injection Alone
Started | 244 | 237
Completed | 244 | 237
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lidocaine Onto Skin Prior to Lidocaine Subcutaneous Injection | Lidocaine Subcutaneous Injection Alone | Total
Number analyzed (Participants) | 244 | 237 | 481
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 58.5 [46.4 to 68.6] | 56.8 [44.8 to 65.4] | 57.4 [45.2 to 67.4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 120 | 105 | 225
  Male | 124 | 132 | 256
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  white, nonhispanic | 136 | 123 | 259
  white, hispanic | 10 | 14 | 24
  african american | 90 | 94 | 184
  asian | 5 | 3 | 8
  other | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Pain Assessment: Overall
Description: Visual analog scale (VAS). This is a standardized analog scale with scores from 0-100. It measures level of pain with 0 meaning no pain and 100 meaning the most extreme level of pain. Higher values refer to a worse outcome.
Time Frame: post procedure (day 1)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lidocaine Onto Skin Prior to Lidocaine Subcutaneous Injection | Lidocaine Subcutaneous Injection Alone
Number analyzed (Participants) | 244 | 237
units on a scale | 15.3 (19.3) | 19.0 (22.8)

2. Secondary Outcome: Pain Assessment: Lidocaine Injection
Description: visual analog scale (VAS) 0= no pain to 100 = worse pain possible
Time Frame: post procedure (day 1)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lidocaine Onto Skin Prior to Lidocaine Subcutaneous Injection | Lidocaine Subcutaneous Injection Alone
Number analyzed (Participants) | 244 | 237
units on a scale | 18.4 (21.2) | 20.8 (23.5)

3. Secondary Outcome: Pain Assessment: During Procedure
Description: visual analog scale (VAS) 0 = no pain to 100 = worse pain possible Rather, this is a pain assessment during the actual procedure rather than during the pre-procedure lidocaine injection.
Time Frame: post procedure (day 1)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lidocaine Onto Skin Prior to Lidocaine Subcutaneous Injection | Lidocaine Subcutaneous Injection Alone
Number analyzed (Participants) | 244 | 237
units on a scale | 12.2 (19.4) | 16.6 (24.8)

ADVERSE EVENTS:
Arm/Group | Lidocaine Onto Skin Prior to Lidocaine Subcutaneous Injection | Lidocaine Subcutaneous Injection Alone
All-Cause Mortality (participants affected / at risk) | 0/244 | 0/237
Serious Adverse Events (participants affected / at risk) | 0/244 | 0/237
Other Adverse Events (participants affected / at risk) | 0/244 | 0/237

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No